CLINICAL TRIAL: NCT00222651
Title: A Phase II Multicenter, Randomized, Double Blind Study Comparing the Efficacy and Safety of Single Bolus i.v. Tenecteplase Versus Placebo in Normotensive Patients With Pulmonary Embolism and Right Ventricular Dysfunction
Brief Title: Tenecteplase Pulmonary Embolism Italian Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: competitor study about to start
Sponsor: University Of Perugia (Other)
Responsible Party: Department of Internal Medicine, University of Perugia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRU-UniPg-01-02
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-04

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; right ventricular dysfunction; thrombolysis; echocardiography
MeSH Terms: conditions — Pulmonary Embolism; Ventricular Dysfunction, Right | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: tenecteplase

SUMMARY:
To assess the efficacy and safety of Tenecteplase versus Placebo in normotensive patients with sub-massive Pulmonary Embolism and Right Ventricular Dysfunction (RVD) all receiving unfractionated heparin (UFH)

DETAILED DESCRIPTION:
In patients with major acute PE thrombolysis has been shown to be life saving (22). Recent registries showed the beneficial effect of thrombolysis also in patients with PE not associated with shock or hypotension (4-23). In these patients thrombolytic treatment has been shown to obtain an improvement of 37% in lung perfusion, detected by lung scan, with respect to an improvement of 18.8% obtained by heparin treatment (24). In a different trial, rt-PA resulted in a faster and greater improvement of pulmonary artery hypertension than heparin treatment (25). Indeed, PE has a wide spectrum of severity at presentation and it is conceivable that the use of more aggressive treatments should be reserved to patients at high risk for adverse outcome. Hence, the search started of prognostic factors of adverse outcome in patients with pulmonary embolism.

RVD has been associated with early adverse outcome (PE recurrence and mortality) in patients with acute PE (26-28; 3). In-hospital mortality in PE patients with and without echocardiographic RVD has been found to be 18.4% and 5.7%, respectively (3). Ribeiro et al. found a higher mortality in patients with PE and severe RVD: in-hospital mortality was 7.9% in the overall population with respect to 14.3% in patients with severe RVD (5). The ICOPER registry reported a 2-week mortality of 15.9% in patients presenting with RVD in comparison with 8% in patients without RVD (23). In MAPPET 10% of patients with RVD died within 30 days as compared to 4.1% of patients without (4).

RVD is a common finding in patients with acute PE and normal blood pressure (BP) (29-33). Recent data suggest that patients with objectively confirmed PE, normal BP and echocardiographic evidence of RVD have a high incidence of adverse outcome (7) and may potentially benefit from more aggressive treatment (34-35). In a recent study patients with acute PE were classified according to the presence of RVD and hypotension; the short-term mortality and the incidence of PE-related shock in patients with normal BP and echo RVD was respectively 5% and 10%. None of the patients with normal BP and no RVD died or experienced PE-related shock (6).

It has been recently demonstrated in patients with PE and pulmonary hypertension or RVD but without arterial hypotension or shock, that rt-PA significantly reduces the incidence of adverse in-hospital outcome events (death and clinical deterioration) with respect to heparin (8).

Consecutive patients with symptomatic PE, since no more than four days, confirmed by objective testing (high probability lung scan or intermediate probability lung scan and objectively confirmed deep vein thrombosis or spiral CT or pulmonary angiography or TE echocardiography) will undergo echocardiographic examination within 24 hour from diagnosis. Patients with RVD and normal BP (Systolic BP> 100 mmHg) will be included in the study.

180 patients will be randomized in the study. The patients included in the study will be randomized, in a double blind fashion, to receive Tenecteplase + UFH (90 patients) or Placebo + UFH (90 patients).

Study treatment should be administered within 6 hours from echocardiography. Echocardiography will be repeated at 24 hours and 7 days or discharge (whichever comes first) from Tenecteplase or Placebo injection. A Follow-up visit at 30 days from randomization will include: clinical history, physical examination and ECG and an echocardiographic examination.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 85;
* symptomatic PE confirmed by: high probability lung scan, or intermediate probability lung scan and objectively confirmed deep vein thrombosis, or spiral CT-scan or pulmonary angiography or TE echocardiography;
* normal blood pressure (SBP >100mmHg);
* RVD at echocardiography (see criteria);
* written informed consent.

Exclusion Criteria:

* absence of RVD at echocardiography;
* shock or hypotension (SBP < 100 mmHg);
* therapeutic heparin (UFH or LMWH) treatment for more than 48 hours prior to randomization;
* administration of thrombolytic agents within the previous 4 days;
* vena cava filter insertion or pulmonary thrombectomy within the previous 4 days
* chronic pulmonary hypertension or severe COPD;
* hypertension defined as blood pressure >180/110 mm Hg (systolic BP >180 mm Hg and/or diastolic BP >110 mm Hg) on a single, reliable measurement during current admission at enrolling site prior to randomisation;
* use of GP IIb/IIIa antagonists within the preceding 7 days;
* significant bleeding disorders either at present or within the past 6 months;
* active peptic ulceration;
* known diabetic haemorrhagic retinopathy or other haemorrhagic ophthalmic conditions;
* known haemorrhagic diathesis;
* known arterial aneurysm and known arterial/venous malformation;
* known neoplasm with increased bleeding risk;
* prolonged cardiopulmonary resuscitation (>10 minutes) in the previous two weeks;
* current oral anticoagulation;
* major surgery, biopsy of a parenchymal organ, or significant trauma within the past 2 months;
* any known history of stroke or transient ischaemic attack (TIA) or dementia;
* any recent head trauma and any other trauma occurring after onset of the current pulmonary embolism;
* any known history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery);
* known subacute bacterial endocarditis;
* known acute pancreatitis;
* known severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension
* (oesophageal varices) and active hepatitis;
* pregnancy or lactation or parturition within the previous 30 days;
* women of childbearing potential must have a negative pregnancy test, or use a medically accepted method of birth control;
* treatment with an investigational drug under another study protocol in the past 7 days;
* previous enrolment in this study;
* known hypersensitivity to Tenecteplase, Alteplase, unfractionated heparin, or to any of the excipients;
* anticipated or obvious problem with vascular access;
* any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated;
* inability to follow protocol requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2004-07; Study Completion 2006-07 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant reduction of RVD | 24 hours from Tenecteplase or Placebo injection

SECONDARY OUTCOMES:
Clinically relevant reduction of RVD; Clinical deterioration requiring escalation of treatment | 7 days from Tenecteplase or Placebo
PE recurrence | 30 days
Death | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Agnelli, MD, Study Chair — Department of Internal Medicine - University of Perugia; Cecilia Becattini, MD, Study Director — Department of Internal Medicine - University of Perugia
Locations (30):
- Italy (30):
  - Dipartimento di Cardiologia - Ospedale del Delta, Lagosanto, Ferrara
  - Unità Operativa di Cardiologia - Azienda Ospedaliera - Ospedale Civile di Vimercate, Desio, Milano
  - Divisione di Cardiologia - Azienda Ospedaliera - Ospedale Civile di Legnano, Legnano, Milano
  - Unità Operativa di Cardiologia - Ospedale di Circolo e Fondazione Macchi, Varese, Milano
  - Divisione Medica II - Ospedale di Vimercate, Vimercate, Milano
  - Medicina D'Urgenza e Pronto Soccorso - Opsedale Regionale, Ancona
  - Divisione di Cardiologia - Azienda Ospedaliera di Venere -Giovanni XXIII, Bari
  - U.O. di Cardiologia - Ospedale di Bentivoglio, Bologna
  - Medicina d'Urgenza - Policlinico S. Orsola, Bologna
  - UTIC - Ospedale Civile di Brescia, Brescia
  - Reparto di Cardiologia - Casa di Cura Poliambulanza - Congregazione Suore Ancelle della Carità, Brescia
  - Medicina D'Urgenza, Cardiologia - Ospedale Civile "San Sebastiano", Caserta
  - Dipartimento di Emergenza Accettazione - Azienda Ospedaliera Universitaria Careggi, Florence
  - Divisione Medica II - Ospedale Galliera, Genova
  - Dipartimento di Emegernza e Accetazione (DEA) - Az. Ospedale-Università San Martino di Genova, Genova
  - Reparto di Cardiologia - Presidio Ospedaliero Piana di Lucca, Lucca
  - Dipartimento Cuore Polmone - Ospedale Carlo Poma, Mantova
  - Reparto di Cardiologia - Azienda Ospedaliera Fatebenfratelli Oftalmico, Milan
  - Medicina D'Urgenza - Ospedale Maggiore Policlinico, Milan
  - Reparto di Pneumologia - Ospedale San Giuseppe, Milan
  - Unità Operativa di Cardiologia - Ospedale S Carlo Borromeo, Milan
  - Medicina D'Urgenza - Az. Osped. Ospedale Niguarda "Cà Granda", Milan
  - Medicina Interna II - Azienda Ospedaliera "Maggiore della Carità" di Novara, Novara
  - Department of Internal Medicine - University of Perugia, Perugia
  - Malattie Apparato Respiratorio - Ospedale Cisanello, Pisa
  - Reparto di Angiologia - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Divisione di Cardiologia - Ospedale Civile, Rovigo
  - Divisione di Pneumologia - Ospedale S Maria, Terni
  - Medicina D'Urgenza - Azienda Ospedaliera S. Giovanni Battista "Le Molinette", Torino
  - Medicina D'Urgenza - Ospedale Cattinara, Trieste

REFERENCES:
- [Derived] Becattini C, Agnelli G, Salvi A, Grifoni S, Pancaldi LG, Enea I, Balsemin F, Campanini M, Ghirarduzzi A, Casazza F; TIPES Study Group. Bolus tenecteplase for right ventricle dysfunction in hemodynamically stable patients with pulmonary embolism. Thromb Res. 2010 Mar;125(3):e82-6. doi: 10.1016/j.thromres.2009.09.017. Epub 2009 Oct 14. PMID 19833379